CLINICAL TRIAL: NCT07146763
Title: A Randomized Trial to Reduce Inappropriate Prescribing to Older Adults Visiting the Emergency Department
Brief Title: A Trial to Reduce Inappropriate Prescribing to Older Adults Visiting the Emergency Department
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2000036876; P30AG024968 (NIH)
Record Dates: First submitted 2025-08-20; First posted 2025-08-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Inappropriate Prescribing
Keywords: Older Adults; Emergency Department; Inappropriate Prescribing
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: The study population are Emergency Medicine prescribers practicing in the Yale New Haven Health System with at least 30 visits with patients over age 65.
  Patients are not target subjects but that their data will be utilized from the medical record, pre- and post-intervention.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Credible Peer Messenger (Experimental): Providers receive automated prescribing feedback messages from a credible peer messenger, including aspirational norms and benchmark comparisons based on Geriatric Emergency Medication Safety Recommendations (GEMS-Rx) recommendations, to promote safer prescribing practices.
  Interventions: Behavioral: Prescribing Feedback
- Anonymous Messenger (Experimental): Providers receive automated prescribing feedback messages from an anonymous messenger system, including aspirational norms and benchmark comparisons based on Geriatric Emergency Medication Safety Recommendations (GEMS-Rx) recommendations, to promote safer prescribing practices.
  Interventions: Behavioral: Prescribing Feedback
- Control group (No Intervention): Providers continue with standard of care. No feedback messages are sent.

INTERVENTIONS:
Behavioral: Prescribing Feedback — Automated prescribing feedback messages are delivered to clinician prescribers in participating emergency departments. Messages are based on Geriatric Emergency Medication Safety Recommendations (GEMS-Rx) recommendations and include aspirational norms and benchmark comparisons. Depending on study arm, feedback is sent either from a credible peer messenger or through an anonymous messenger system.
  Arms: Anonymous Messenger; Credible Peer Messenger

SUMMARY:
Cluster-randomized trial assessing the impact of interventions on guideline-concordant prescribing in Emergency Departments (ED). The study compares the effectiveness of feedback messages about potentially inappropriate medications (PIMs) delivered by peer clinician prescribers or anonymous systems, compared to standard of care. The goal is to reduce PIM prescribing for older adults discharged from emergency departments.

DETAILED DESCRIPTION:
The goal of this trial is to compare the effectiveness of prescribing feedback delivered by a credible peer messenger and by an anonymous messaging system against standard of care in emergency departments. This intervention to Emergency Department (ED) clinician prescribers is a modification of previous studies that optimizes feedback about Potentially Inappropriate Medications (PIMs) using findings from behavioral science. Clinician prescribers who meet eligibility criteria and provide digital affirmative consent will be enrolled if they have encounters in a participating ED facility. The Joint Data Analytics Team (JDAT) will identify patients aged 65 years and older who were seen in the ED to evaluate prescribing outcomes. The focus of this registration is the randomized trial.

ELIGIBILITY:
Inclusion Criteria:

1. Licensed clinicians with prescribing authority (physician, advanced practice registered nurse, or physician assistant)
2. Practicing in one of the participating Yale New Haven Health System emergency departments
3. At least 30 Emergency Department (ED) discharge encounters with patients aged 65 years or older in the 12 months preceding study enrollment
4. Provides digital affirmative consent to participate

Exclusion Criteria:

* Failure to meet inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change PIM prescribing rate | At ED discharge, calculated monthly, using rolling 90-day prescribing data, over the 12-month intervention period and 6-month follow-up
  Change in potentially inappropriate medication (PIM) prescribing rate based on the Geriatric Emergency Medication Safety Recommendations (GEMS-Rx). Outcome is measured as the percentage of Emergency Department (ED) discharge prescriptions for PIMs among patients aged 65 years or older.

SECONDARY OUTCOMES:
Changes in prescribing by medication class | At ED discharge, calculated monthly, using rolling 90-day prescribing data, over the 12-month intervention period and 6-month follow-up
  Changes in prescribing rates for high-risk medication classes identified in the GEMS-Rx based on percentage of ED discharge prescriptions for each targeted medication class among patients aged 65 years or older.
Adoption of alternative recommendations | Monthly during the 12-month intervention period and 6-month follow-up
  Percentage of ED discharge encounters in which a recommended alternative medication was prescribed in place of a PIM based on percentage of eligible encounters.
Access to Epic workbench reports | Monthly during the 12-month intervention period and 6-month follow-up
  Access to Epic workbench prescribing reports and message links (including Frequently Asked Questions, FAQs) based on number of accesses per clinician per month.
Mean overall readmission rate | Measured at 30 days post-discharge for all eligible ED visits during the 12-month intervention period and 6-month follow-up
  All-cause readmission rates will be monitored to assess safety based on percentage of ED discharge encounters followed by any hospital readmission within 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Daniella Meeker, PhD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital Emergency Departments, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be transferred to the National Archive for Computerized Data On Aging (NACDA)
Time Frame: Made available upon publication.